CLINICAL TRIAL: NCT03881553
Title: Interventions to Help Infants and Children Recover in the Hospital
Brief Title: Interventions to Help Infants Recover in the Hospital
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid halt in March; PI moved to another Institution
Sponsor: Elisabeth Salisbury, PhD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Elisabeth Salisbury, PhD, Research Associate Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H00015487; U54HL143541 (NIH)
Record Dates: First submitted 2019-03-03; First posted 2019-03-19 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Infant Apnea; Neonatal Abstinence Syndrome; Sleep
Keywords: Prematurity; Neonatal Abstinence Syndrome; Autonomic Function; Sleep; Stochastic Resonance; Newborn/Infant
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Premature Birth

STUDY DESIGN:
Intervention Model Description: Within-subjects design. Each subject will serve as own control and receive periods of intervention and no intervention within a study session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Premature Infants (NICU) (Experimental): Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) will participate in up to 2 sessions with NEATCAP intervention and up to 2 sessions with SVS mattress intervention.
  Interventions: Device: NEATCAP; Device: SVS mattress
- Opioid-Exposed Newborns (NICU) (Experimental): Opioid-exposed newborns receiving care in the Neonatal Intensive Care Unit (NICU) will participate in up to 2 sessions with NEATCAP intervention and up to 2 sessions with SVS mattress intervention.
  Interventions: Device: NEATCAP; Device: SVS mattress
- Hospitalized Infants (PICU) (Experimental): Infants receiving treatment in the Pediatric Intensive Care or Inpatient Unit will participate in up to 2 sessions with NEATCAP intervention and up to 2 sessions with SVS mattress intervention.
  Interventions: Device: NEATCAP; Device: SVS mattress

INTERVENTIONS:
Device: NEATCAP — NEATCAP: Neurosensory, Environmental Adaptive Technology is a sound attenuating earmuff that reduces unsafe high-frequency noise.
  Other Names: NEATCAP DREAMIES (NEATCap Medical, LLC)
Device: SVS mattress — SVS mattress: Stochastic Vibratory Stimulation is a mattress that provides gentle, random, vibrotactile stimulation.

SUMMARY:
This pilot project will evaluate independently two non-pharmacological interventions, 1) Neurosensory, Environmental Adaptive Technology (NEATCAP) and 2) Stochastic Vibrotactile Stimulation (SVS), as adjuvant non-pharmacological interventions for improving sleep and cardio-respiratory function in hospitalized infants. Within-subject design allows subjects to serve as their own control and receive periods of routine care with and without intervention. One intervention will be evaluated per study session. Infants may participate in up to four sessions.

DETAILED DESCRIPTION:
Infants and children treated in the hospital often present with autonomic and sleep disturbances that may be related to prematurity, opioid and other drug exposures in utero, illness, surgery, medical procedures, and/or treatment medications. In addition, patients treated in neonatal and pediatric units often require prolonged hospitalization with medical monitoring and life-sustaining devices equipped with patient safety alarms. Such bedside equipment may result in patients being exposed to loud and/or persistent noises that may further disrupt sleep and autonomic function and compromise recovery and outcomes.

This pilot study will study three separate pediatric populations being treated in neonatal and pediatric hospital units: 1) Premature Infants; 2) Opioid-exposed newborns requiring medication for Neonatal Abstinence Syndrome; and 3) Hospitalized infants treated for illness or surgery. Subjects will participate in up to 4 study sessions during their hospitalization, testing independent effects of two interventions complementary to routine care: 1) Neurosensory, Environmental Adaptive Technology (NEATCAP), and 2) stochastic vibrotactile stimulation (SVS). Within-subject design will allow for comparisons between periods, i.e., with and without the study-session intervention, separately for each device, for improving sleep and cardio-respiratory function in three independent groups of hospitalized infants.

ELIGIBILITY:
Inclusion Criteria:

* Pre-term infants (>30 wks PMA) and full-term newborns receiving care since birth in the NICU/CCN.
* Infants/Children receiving care in the PICU/PIU (may have had a history of prematurity).
* May be with or without in utero opioid exposure and/or other drug exposure (prescribed or illicit).
* May have received or be receiving opioids and/or other treatment medications as part of their medical-care plan.
* Infants and children on respiratory support and/or with medical complications will not be excluded if these complications are potentially reversible.

Exclusion Criteria:

* Congenital anomalies of the head and/or neck.
* Significant cranial trauma.
* Hydrocephalus.
* Current or history of intraventricular hemorrhage>grade 2.
* Clinically significant cardiac shunt.
* Hemodynamic instability requiring pharmacological intervention at time of study participation.
* Documented HIV and/or MRSA positivity requiring treatment at time of study participation.
* Seizure disorder not due to opioid withdrawal.
* Invasive ventilation at time of study participation.
* Recommendation of attending physician or primary medical caregiver not to enroll the patient for any reason.

Ages: 2 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Salisbury, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuzarte I, Indic P, Barton B, Paydarfar D, Bednarek F, Bloch-Salisbury E. Vibrotactile stimulation: A non-pharmacological intervention for opioid-exposed newborns. PLoS One. 2017 Apr 20;12(4):e0175981. doi: 10.1371/journal.pone.0175981. eCollection 2017. PMID 28426726
- [Background] Bloch-Salisbury E, Indic P, Bednarek F, Paydarfar D. Stabilizing immature breathing patterns of preterm infants using stochastic mechanosensory stimulation. J Appl Physiol (1985). 2009 Oct;107(4):1017-27. doi: 10.1152/japplphysiol.00058.2009. Epub 2009 Jul 16. PMID 19608934
- [Background] Balsan MJ, Burns J, Kimock F, Hirsch E, Unger A, Telesco R, Bloch-Salisbury E. A pilot study to assess the safety, efficacy and ease of use of a novel hearing protection device for hospitalized neonates. Early Hum Dev. 2021 May;156:105365. doi: 10.1016/j.earlhumdev.2021.105365. Epub 2021 Mar 26. PMID 33857731
- [Result] Bloch-Salisbury E, McKenna L, Boland E, Chin D. Assessment of a hearing protection device on infant sleep in the neonatal intensive care unit. J Sleep Res. 2023 Apr;32(2):e13610. doi: 10.1111/jsr.13610. Epub 2022 Apr 22. PMID 35460141
- See also: A Pilot Study to Evaluate Patient Tolerance and Nursing Ease-of-Use of a Novel Hearing Protection Device (NEATCAP) — https://clinicaltrials.gov/ct2/show/NCT02744066?term=neatcap&rank=1
- See also: Efficacy and Outcomes of a Non-Pharmacological Intervention for Neonatal Abstinence Syndrome — https://clinicaltrials.gov/ct2/show/NCT02801331?term=Salisbury&cond=NAS&rank=2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in the neonatal and pediatric hospital units where infants receiving in-patient care.
Pre-assignment Details: Within-subject design so each participant received periods with and without the intervention (NEATCAP and SVS mattress device). Assignment was based on equipment availability. Number of study sessions may have been related to: discharged from hospital prior to opportunity to participate in 1 or more study sessions; i.e., personnel and/or equipment availability to schedule session; Covid-19 halt on in-person subject participation; termination of project.
Groups:
- Premature Infants (NICU): Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) participated in 1 session with NEATCAP.
- Opioid-Exposed Newborns (NICU): Opioid-exposed newborns receiving care in the Neonatal Intensive Care Unit (NICU) participated in 1 session with NEATCAP.
- Hospitalized Infants (PICU): Infants receiving treatment in the Pediatric Intensive Care or Inpatient Unit participated in up to 2 sessions with SVS mattress intervention.
Period: Overall Study
Arm/Group | Premature Infants (NICU) | Opioid-Exposed Newborns (NICU) | Hospitalized Infants (PICU)
Started | 11 | 2 | 4
Completed | 10 | 1 | 3
Not Completed | 1 | 1 | 1
Not completed — Discharged prior to participation | 1 | 1 | 0
Not completed — Developed infection prior to participation--excluded per protocol criteria | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Reported only on Arm 1 infants who participated in the study session. Did not report on participants in Arm 2 or Arm 3 due to small number of participants risk of potential identification.
  Data not collected on enrolled (consented) who did not participate in the study intervention.
Groups:
- Experimental: Premature Infants (NICU): Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) will participate in up to 2 sessions with NEATCAP intervention and up to 2 sessions with SVS mattress intervention.
- Experimental: Opioid-Exposed Newborns (NICU): Opioid-exposed newborns receiving care in the Neonatal Intensive Care Unit (NICU) will participate in up to 2 sessions with NEATCAP intervention and up to 2 sessions with SVS mattress intervention.
- Experimental: Hospitalized Infants (PICU): Infants receiving treatment in the Pediatric Intensive Care or Inpatient Unit will participate in up to 2 sessions with NEATCAP intervention and up to to 2 sessions with SVS mattress intervention.
- Total: Total of all reporting groups
Arm/Group | Experimental: Premature Infants (NICU) | Experimental: Opioid-Exposed Newborns (NICU) | Experimental: Hospitalized Infants (PICU) | Total
Number analyzed (Participants) | 10 | 2 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: Count of participants includes only those subjects who participated in the study intervention. Data was not collected on enrolled (consented) subjects who did not participate in study intervention (i.e., discharged or withdrawn prior to any data collection).
  Participants
    number analyzed (Participants) | 10 | 1 | 3 | 14
    <=18 years | 10 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Population: Count of participants includes only those subjects who participated in the study intervention. Data was not collected on enrolled (consented) subjects who did not participate in study intervention (i.e., discharged or withdrawn prior to any data collection).
  weeks
    Mean Gestational Age (weeks): number analyzed (Participants) | 10 | 1 | 3 | 14
    Mean Gestational Age (weeks) | 34.1 (1.3) | NA (NA) — Due to small n, risk of potential identification | NA (NA) — Due to small n, risk of potential identification | NA (NA) — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Count of participants includes only those subjects who participated in the study intervention. Data was not collected on enrolled (consented) subjects who did not participate in study intervention (i.e., discharged or withdrawn prior to any data collection).
  Participants
    number analyzed (Participants) | 10 | 1 | 3 | 14
    Female | 5 | NA — Due to small n, potential risk of participant identification | NA — Due to small n, potential risk of participant identification | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | 5 | NA — Due to small n, potential risk of participant identification | NA — Due to small n, potential risk of participant identification | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Count of participants includes only those subjects who participated in the study intervention. Data was not collected on enrolled (consented) subjects who did not participate in study intervention (i.e., discharged or withdrawn prior to any data collection).
  Participants
    number analyzed (Participants) | 10 | 1 | 3 | 14
    Hispanic or Latino | 3 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Not Hispanic or Latino | 7 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Unknown or Not Reported | 0 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Count of participants includes only those subjects who participated in the study intervention. Data was not collected on enrolled (consented) subjects who did not participate in study intervention (i.e., discharged or withdrawn prior to any data collection).
  Participants
    American Indian or Alaska Native | 0 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Asian | 0 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Native Hawaiian or Other Pacific Islander | 0 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Black or African American | 0 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    White | 6 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    More than one race | 1 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Unknown or Not Reported | 3 | NA — Due to small n, potential risk of participant identification. | NA — Due to small n, potential risk of participant identification. | NA — Total not calculated because data are not available (NA) in one or more arms.
Mean Post-Menstrual Age at time of 1st session [Mean (Standard Deviation); unit: weeks] — Population: Count of participants includes only those subjects who participated in the study intervention. Data was not collected on enrolled (consented) subjects who did not participate in study intervention (i.e., discharged or withdrawn prior to any data collection).
  weeks | 35.84 (1.2) | NA (NA) — Due to small n, potential risk of participant identification. | NA (NA) — Due to small n, potential risk of participant identification. | NA (NA) — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Sleep Rate With and Without NEATCAP Intervention
Description: Within each Group, percent sleep (and inversely percent wake) duration will be compared for periods of device on and device off separately for each intervention device within each study session.
Time Frame: Between 8 to 12 hours (reflecting 3 interfeed periods NEATCAP OFF then ON then OFF)
Measure: Mean (Standard Deviation); unit: percent of period sleep
Groups:
- Premature Infants (NICU): Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) participated in 1 session with NEATCAP intervention
  NEATCAP: NEATCAP: Neurosensory, Environmental Adaptive Technology is a sound attenuating earmuff that reduces unsafe high-frequency noise.
Arm/Group | Premature Infants (NICU)
Number analyzed (Participants) | 10
percent of period sleep
  NEATCAP OFF1 | 79.99 (19.49)
  NEATCAP ON | 94.11 (9.07)
  NEATCAP OFF2 | 75.74 (25.46)
Statistical Analysis 1: Comparison: Premature Infants (NICU); Test type: Other — Non-parametric Friedmans; p = 0.081, Friedman's — χ2 =5.03
Statistical Analysis 2: Comparison: Premature Infants (NICU); Test type: Other — Post hoc: Wilcoxon; p = 0.05, Wilcoxon (Mann-Whitney) — ON1 compared to OFF1
Statistical Analysis 3: Comparison: Premature Infants (NICU); Test type: Other — Post Hoc Wilcoxon; p = 0.021, Wilcoxon (Mann-Whitney) — ON1 compared to OFF2

2. Primary Outcome: Mean Respiratory Rate With and Without Intervention
Description: Within each Group, mean respiratory rate will be compared for periods of device on and device off separately for each intervention device within each study session.
Time Frame: Between 8 to 12 hours (reflecting 3 interfeed periods NEATCAP OFF then ON then OFF)
Measure: Mean (Standard Deviation); unit: breaths/min
Groups:
- Premature Infants (NICU): Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) participated in 1 session with NEATCAP intervention
  NEATCAP: NEATCAP: Neurosensory, Environmental Adaptive Technology is a sound attenuating earmuff that reduces unsafe high-frequency noise.
  .
Arm/Group | Premature Infants (NICU)
Number analyzed (Participants) | 10
breaths/min
  Respiratory Rate OFF1 | 66.7 (13.6)
  Respiratory Rate ON | 62.6 (8.2)
  Respiratory Rate OFF2 | 64.9 (10.9)

3. Primary Outcome: Mean Heart Rate With and Without Intervention
Description: Within each Group, mean heart rate will be compared for periods of device on and device off separately for each intervention device within each study session.
Time Frame: Between 8 to 12 hours (reflecting 3 interfeed periods NEATCAP OFF then ON then OFF)
Measure: Mean (Standard Deviation); unit: beats/min
Groups:
- Premature Infants (NICU): Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) w participated in 1 session with NEATCAP intervention
  NEATCAP: NEATCAP: Neurosensory, Environmental Adaptive Technology is a sound attenuating earmuff that reduces unsafe high-frequency noise.
Arm/Group | Premature Infants (NICU)
Number analyzed (Participants) | 10
beats/min
  Heart Rate OFF1 | 149.8 (13.5)
  Heart Rate ON | 151.8 (13.4)
  Heart Rate OFF2 | 149.6 (12.9)

4. Secondary Outcome: Mean Movement Activity
Description: Within each Group, mean movement activity will be compared for periods of device on and device off separately for each intervention device within each study session.
Time Frame: Between 8 to 12 hours (reflecting 3 interfeed periods NEATCAP OFF then ON then OFF)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Premature Infants (NICU)
Number analyzed (Participants) | 10
percent
  Percent Movement OFF1 | 26.4 (6.8)
  Percent Movement ON | 26.9 (8.6)
  Percent Movement OFF2 | 33.2 (7.0)

ADVERSE EVENTS:
Time Frame: up to 24 hours following completion of a study session
Description: Potential risk of adverse events described in IRB study plan and consent form include: skin irritation and or rash due to NEATCAP device and/or additional sensors used to record physiological signals that does not resolve by end of study session. Subsequent report by bedside medical caregiver of exacerbated function post study session not apparently related to infant current problems.
Groups:
- Premature Infants (NICU): NEATCAP Device: Premature infants receiving care in the Neonatal Intensive Care Unit (NICU) will participated in 1 session with NEATCAP intervention
- Opioid-Exposed Newborns (NICU): NEATCAP Device: Opioid-exposed newborns receiving care in the Neonatal Intensive Care Unit (NICU) participate in 1 session with NEATCAP intervention.
- Hospitalized Infants (PICU): Mattress Device: Infants receiving treatment in the Pediatric Intensive Care participate in up to 2 sessions with SVS mattress intervention.
Arm/Group | Premature Infants (NICU): NEATCAP Device | Opioid-Exposed Newborns (NICU): NEATCAP Device | Hospitalized Infants (PICU): Mattress Device
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/1 | 0/3

LIMITATIONS AND CAVEATS:
Early termination leading to incomplete arms of trial. Accordingly, due to small n from the early termination of the trial, outcomes in Arm 2 and Arm 3 are not reported due to potential risk of participant identification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03881553/Prot_SAP_001.pdf